CLINICAL TRIAL: NCT05759039
Title: A Randomized Clinical Pilot Trial Comparing Isolated Medial Patellofemoral Ligament Reconstruction to Medial Patellofemoral Ligament Reconstruction Combined with Tibial Tubercle Osteotomy: SHould You TransFer the Tubercle (SHYFT)?
Brief Title: SHould You TransFer the Tubercle?
Acronym: SHYFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Banff Sport Medicine Foundation (Other)
Collaborators: Canadian Orthopaedic Foundation (Other); CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB17-1256
Record Dates: First submitted 2023-02-17; First posted 2023-03-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Patellofemoral Dislocation; Tibial Tubercle Osteotomy; Medial Patellofemoral Ligament Reconstruction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MPFL-R (Active Comparator): Medial patellofemoral ligament reconstruction
  Interventions: Procedure: Medial patellofemoral ligament reconstruction
- MPFL-R + TTO (Active Comparator): Medial patellofemoral ligament reconstruction with concomitant tibial tubercle osteotomy
  Interventions: Procedure: Medial patellofemoral ligament reconstruction; Procedure: Tibial tubercle osteotomy

INTERVENTIONS:
Procedure: Medial patellofemoral ligament reconstruction — Medial patellofemoral ligament reconstruction
Procedure: Tibial tubercle osteotomy — Tibial tubercle osteotomy
  Arms: MPFL-R + TTO

SUMMARY:
The aim of this study is to investigate the role of tibial tubercle osteotomy (TTO) on the subjective and objective outcomes following medial patellofemoral ligament reconstruction (MPFL-R) in patients with an increased tibial tubercle-trochlear groove (TT-TG) distance with or without patella alta.

This Pilot RCT will assess the feasibility of conducting this study for:

1. The ability to recruit study patients
2. Adherence to the study protocol
3. Completion rates of patient follow-up at a minimum of 12 months post-operative

DETAILED DESCRIPTION:
For patients with recurrent lateral patellofemoral instability, a medial patellofemoral ligament reconstruction (MPFL-R) consistently provides significant improvements in symptoms, quality of life, and return to sport. During an MPFL-R the surgeon will place a soft tissue graft from the medial patella to the femur. The graft used to create the new MPFL can be autograft (usually hamstring tendon) or allograft.

The tibial tubercle osteotomy (TTO) is a procedure designed to change the vector of the pull of the quadricep muscles by moving the insertion point of the patellar tendon. This is achieved by transferring the tendon with a block of bone to allow for consistent and reliable healing. The TTO is a versatile procedure that can move the patellar tendon insertion medially, anteriorly, or distally, or a combination of these directions. It can be used to correct a lateralized tibial tubercle or patella alta.

Despite the association of an increased TT-TG distance with patellofemoral instability, it has been difficult to demonstrate a correlation with patient outcomes after patellar stabilisation surgery. In addition, studies have been unable to correlate the pre-operative presence of patella alta with clinical outcomes after MPFL-R.

This randomized clinical pilot trial will randomly allocate patients with lateral patellofemoral instability and an elevated TT-TG distance with or without patella alta ato receive either an isolated MPFL-R or an MPFL-R in combination with a correcting TTO (medializing, distalizing, or a combination of both).

Patients will be followed for two years post-operative with subjective outcome measures and objective clinical and functional testing.

The study groups will be:

1. Isolated MPFL-R
2. MPFL-R with a TTO

The primary outcome measures will be:

1. Number of study patients recruited
2. Adherence to the study protocol (number of protocol deviations)
3. Follow-up completion rates of study patients at a minimum of 12 months post-operative

Secondary outcome measures include the Banff Patellar Instability Instrument 2.0 (BPII 2.0), functional testing, clinical assessment, complications, re-dislocation rate, post-operative pain scores, patient satisfaction, and patient-reported outcome scores.

If feasibility is demonstrated via this Pilot RCT, a larger RCT will be designed to answer important questions on how to optimize outcomes and limit morbidity after MPFL-R.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-30 years
* Symptomatic recurrent lateral patellofemoral instability
* TT-TG ≥15mm measured on MRI or ≥18mm on CT scan
* Closed physes (confirmed on knee x-rays)

Exclusion Criteria:

* Caton-Deschamps ratio ≥ 1.4 on lateral radiographs
* Femoral anteversion ≥ 25 degrees on diagnostic imaging rotational profile
* Tibial external rotation ≥ 45 degrees on diagnostic imaging rotational profile
* High-grade trochlear dysplasia requiring trochleoplasty
* Significant osteoarthritis on skyline plain imaging (Kellgren Lawrence grade ≥ 2)
* A chondral lesion of the patellofemoral joint that is undergoing a cartilage restoration procedure.
* Unable to complete computer-based outcome questionnaires
* Pregnant (at time of surgery)

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility - patient recruitment | 12-months post-operative
  Number of study patients recruited
Study Feasibility - protocol adherence | 12-months post-operative
  Adherence to the study protocol (total number of protocol deviations)
Study Feasibility - follow-up completion | 12-months post-operative
  Number of patients completing follow-up a minimum of 12 months post-operative

SECONDARY OUTCOMES:
Banff Patellofemoral Instability Instrument (BPII 2.0) | Baseline, and 6-,12- & 24-months post-operative
  Disease-specific patient-reported outcome measure that assesses quality of life across 5 domains. Scored out of 100, with 100 representing the maximum score for disease-specific quality of life.
Functional Outcomes - Hop Testing | 6-, 12- & 24-months post-operative
  Limb Symmetry Index on 4 single-leg hop test battery (assessed as percentage score operative / non-operative limb)
Patellar Apprehension Test | 6-, 12- & 24-months post-operative
  Rate of positive patellar apprehension
Complications | 6-, 12- & 24-months post-operative
  Rate of post-operative complications including infection, blood clots, reduced range of motion, persistent pain, persistent swelling, and re-dislocations
Post-operative Knee Pain | 6-, 12- & 24-months post-operative
  Post-operative pain score measured on a 10-point visual analogue scale
  The Pain VAS is anchored by 0, which corresponds to "no pain", and 10, which corresponds to the "worst possible pain".
Patient satisfaction | 12- & 24-months post-operative
  Measured on a 5-point Likert scale
  A 5-point patient satisfaction scale measures patient happiness with healthcare services, ranging from 5 (very satisfied) to 1 (very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Hiemstra, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Banff Sport Medicine, Canmore, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No